CLINICAL TRIAL: NCT04890795
Title: A Single Arm, Open, Non Randomized, Phase Ib / IIA Study to Evaluate the Safety and Preliminary Efficacy of AL8326 in the Treatment of Small Cell Lung Cancer
Brief Title: A Phase Ib / IIA Study of AL8326 in Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Advenchen Laboratories Nanjing Ltd. (Industry)
Responsible Party: Sponsor
Organization: Advenchen Laboratories, LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL8326-CN-004
Record Dates: First submitted 2021-04-26; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AL8326 (Experimental): Subject will received AL8326 once daily for 28-days cycle until intolerable toxicity or disease progression or death or voluntary withdrawal the end of this study.During treatment, subjects will be evaluated for anti-tumor efficacy and corresponding safety examinations every 2 cycles, and tumor disease status will be according to RECIST 1.1.
  Interventions: Drug: AL8326 tablets

INTERVENTIONS:
Drug: AL8326 tablets — 10mg/tablet;Oral administration, once daily.
  Other Names: AL8326

SUMMARY:
Based on indicators such as 24 week progression free survival (24 weeks PFS) in small cell lung cancer (SCLC) patients without disease progression after first-line platinum containing chemotherapy, objective response rate (ORR) in SCLC patients with recurrence or progression after first-line platinum containing chemotherapy, and orr in SCLC patients with recurrence or progression after second-line and above treatment,Evaluation of the effectiveness of al8326 monotherapy in small cell lung cancer.

DETAILED DESCRIPTION:
This trial is a multicenter, single arm, open label, nonrandomized, phase Ib / IIA trial that will evaluate the preliminary efficacy and safety of AL8326 in patients with small cell lung cancer (SCLC).Three treatment groups were used in this trial, and the study population, sample size, and basic design of each group were as follows:

Group A: Patients with small-cell lung cancer without disease progression (in remission [PR or Cr] or stable disease [SD] status) after first-line platinum containing chemotherapy were included, with a total sample size expected to be 79 patients.

Group B: Patients who relapsed or progressed after first-line platinum containing chemotherapy regimens, with a total sample size expected to be 79 patients.

Group C: Patients with small cell lung cancer who have relapsed or progressed after at least one line of treatment (including first-line platinum containing therapy, second-line single agent or other) with a total sample size expected to be 79 patients.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects or legal surrogates were required to give written, ethics committee approved informed consent prior to initiation of any screening procedures;
2. Age ≥ 18 years, both genders, patients with histologically confirmed SCLC, and fulfilling the following criteria:

   Group A: Patients with small-cell lung cancer without disease progression (in remission [PR or Cr] or stable disease [SD] status according to RECIST 1.1 criteria) after first-line platinum containing chemotherapy, including extensive stage and limited stage who were not eligible for radical radiotherapy, received four to six cycles of platinum containing chemotherapy previously; Group B: Patients with small-cell lung cancer who have relapsed or progressed after first-line platinum containing chemotherapy regimens; Group C: Patients with small cell lung cancer who have relapsed or progressed after at least one line of therapy (including first-line platinum containing therapy, second-line single agent therapy, or other);Notes: platinum containing chemotherapy regimens included etoposide + cisplatin, etoposide + carboplatin, irinotecan + cisplatin, irinotecan + carboplatin, etoposide + lobaplatin;Second line monotherapy regimens include topotecan, irinotecan, paclitaxel, docetaxel, gemcitabine, oral etoposide, vinorelbine, temozolomide, ifosfamide;Second line and beyond other treatments include small molecule targeted agents, monoclonal antibodies, etc.
3. ECOG (PS) score was 0,1;
4. Life expectancy ≥ 12 weeks;
5. Subjects in arm B / C had at least one measurable tumor lesion according to response evaluation criteria in solid tumors (RECIST 1.1;
6. The subject had adequate organ and bone marrow function meeting the following laboratory test criteria:

   1. Bone marrow function: absolute neutrophil count (ANC) ≥ 1.5×10^9 / L (1500 / mm^3), platelets ≥ 80×10^9/L;
   2. Hemoglobin ≥ 9.0 g / dl;Liver function: serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN), with the exception of patients with Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that manifests as elevated unconjugated bilirubin in the absence of evidence of hemolysis or liver pathology);
   3. Those without liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN, those with liver metastases, ALT and AST ≤ 5×ULN;
   4. Renal function: serum creatinine ≤ 1.5×ULN and a standard endogenous creatinine clearance ≥ 60 ml / min estimated by the Cockcroft Gault formula, CCR (ml / min) = [(140 - age)×Weight (kg)] / [72× SCR (mg / dl)], females as calculated×0.85;
   5. Coagulopathy: international normalized ratio (INR) ≤ 1.5;
   6. Hemodynamically stable and left ventricular ejection fraction (LVEF) ≥ 50% as determined by echocardiography;
7. Previous treatment with cytotoxic chemotherapy, traditional Chinese medicine, ending at least 4 weeks apart from first dose, receipt of nitroso or mitomycin at least 6 weeks apart, and TKI class molecularly targeted agents at least 4 weeks apart and having recovered to grade ≤ 1 from the toxic effects of previous chemotherapy, with the following exceptions: a.alopecia;b. Long term toxicity caused by radiotherapy, which could not be recovered after the judgment of the investigator;c. Platinum induced grade 2 and the following neurotoxicity such as hearing impairment (according to common terminology criteria for adverse events CTCAE V5.0);
8. Women of childbearing age and all male subjects must agree to use highly effective methods of contraception (condoms, contraceptive sponges, contraceptive gels, contraceptive membranes, IUDs, oral or injectable contraceptives, subcutaneous implants, etc.) for the duration of the study and for 3 months after discontinuation.

Exclusion Criteria:

1. Patients who had used AL8326 tablets in the past;
2. Allergic to AL8326 or its analogues, or to any component in the prescription of AL8326;
3. The patients with leptomeningeal history or leptomeningeal metastasis or central nervous system (CNS) metastasis at the time of screening had uncontrollable brain metastasis, spinal cord compression and cancerous meningitis within 8 weeks after the first medication, Patients with CNS metastasis or spinal cord compression whose clinical status is stable and does not need corticosteroid treatment and whose screening time is more than 4 weeks before treatment (including radiotherapy or surgery) are excluded;
4. Patients with current or previous second tumor (except for fully treated basal cell carcinoma of skin or squamous cell carcinoma, cervical carcinoma in situ), unless radical treatment has been carried out and there is no evidence of recurrence and metastasis in the past 5 years;
5. Those who have obvious gastrointestinal history or current diseases, such as inability to swallow, severe peptic ulcer, uncontrollable nausea and vomiting, chronic diarrhea, intestinal obstruction or other chronic gastrointestinal diseases that are difficult to control in recent 3 months, inability to swallow drugs or may affect the intake, transportation or absorption of drugs, or who have undergone total gastrectomy before;
6. Patients with other important primary diseases, such as single drug uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and / or diastolic blood pressure ≥ 100 mmHg), arrhythmias that need clinical intervention (such as long QT syndrome, unmeasurable bazetts corrected QTc or male > 450 ms, female > 470 MS), abnormally prolonged arrhythmias caused by unstable coronary artery disease Patients with decompensated congestive heart failure (NYHA grade III or IV) or myocardial infarction, grade 2 or above thyroid disease, ascites or uncontrolled pleural effusion (CTCAE 5.0 ≥ 2), history of thrombosis or stroke, autoimmune disease, and mental illness within 6 months before administration of the test drug;
7. The patients with arteriovenous thrombotic events such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism in the first 6 months were screened;
8. The tumor had invaded the important blood vessels or the researchers judged that the tumor was likely to invade the important blood vessels during the follow-up study and cause fatal massive hemorrhage;
9. Uncontrolled infection (within 2 weeks before the administration of the test drug);
10. Urine routine examination showed that urine protein was ≥ + +, and 24-hour urine protein was more than 1.0 G;
11. The patients with grade 1 or more bleeding events (according to CTCAE 5.0 > grade 1), including gastrointestinal tract, respiratory system, tumor, urinary tract and cerebral hemorrhage, were screened;
12. Patients treated with anticoagulants or vitamin K antagonists (such as warfarin, heparin or their analogues); Under the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, it is allowed to use low-dose anticoagulants for preventive purposes, such as warfarin (not more than 1 mg daily, oral), low-dose heparin (not more than 12000 u daily) or low-dose aspirin (not more than 100 mg daily);
13. Hepatitis C virus (HCV) antibody, Treponema pallidum antibody or human immunodeficiency virus (HIV) antibody test results of any one or more positive, or active hepatitis B patients (defined as HBV DNA ≥ 2000 IU / ml or HBV DNA ≥ 104 copies);
14. Patients who received any trial drug treatment within 30 days before signing the informed consent form;
15. Patients who received red blood cell or platelet transfusion within 14 days before the first administration;
16. Received major surgical treatment within 4 weeks before signing the informed consent (the patient must fully recover and stabilize before the start of treatment);
17. Patients with previous organ transplantation history or preparing for organ transplantation;
18. Pregnant or lactating female patients;
19. According to the judgment of the investigator, there are other reasons that are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
(Group A) 24 weeks progression free survival (24 weeks PFS) | Every 2 cycles(each cycle is 28--days)
  Objective to evaluate the 24 week progression free survival (24 weeks PFS) of AL8326 in patients with small cell lung cancer (SCLC) without disease progression (PR or CR or SD) after first-line platinum based chemotherapy.
(Group B and C) Objective response rate (ORR) | Every 2 cycles(each cycle is 28--days)
  Objective response rate (ORR) of SCLC patients with recurrence or progression after first-line platinum chemotherapy, and objective response rate (ORR) of SCLC patients with recurrence or progression after second-line or above treatment.

SECONDARY OUTCOMES:
Safety and tolerance(Number of participants with treatment-related adverse events as assessed by CTCAE v5.0) | Every 2 cycles(each cycle is 28--days)
  Objective to evaluate the safety and tolerability of al8326 monotherapy in patients with small cell lung cancer (SCLC) without disease progression (PR or CR or SD) after first-line platinum based chemotherapy; Safety and tolerability in patients with small cell lung cancer who relapsed or progressed after first-line platinum based chemotherapy; Safety and tolerability in patients with small cell lung cancer who relapse or progress after at least second-line treatment (including first-line platinum containing therapy, second-line monotherapy or other treatments).

CONTACTS AND LOCATIONS:
Overall Officials: xiaochun Zhang, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (9):
- China (9):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang